CLINICAL TRIAL: NCT02303600
Title: Fractional Concentration of Exhaled NO(FENO) to Direct Montelukast Treatment of Sub-acute Cough:A Prospective, Open Label, Randomized and Placebo-Controlled Trial
Brief Title: Fractional Concentration of Exhaled NO(FENO) to Direct Montelukast Treatment of Sub-acute Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Min Liu, resident, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAC2014
Record Dates: First submitted 2014-11-17; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Coughing
Keywords: Sub-acute cough
MeSH Terms: conditions — Cough | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- biomarker treatment arm (Experimental): Patients in biomarker guided positive treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) . Patients in biomarker guided negative treatment arm were given placebo tablets (main excipient lactose monohydrate).
  Interventions: Other: Placebo
- standard treatment arm (Active Comparator): Patients in standard treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) .
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Patients in biomarker guided positive treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.). Patients in biomarker guided negative treatment arm were given placebo tablets . Patients in standard treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) . All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.
  Arms: standard treatment arm
Other: Placebo — Patients in biomarker guided negative treatment arm were given placebo tablets (main excipient lactose monohydrate) (p.o., 10mg, q.d.) .
  Other Names: Placebo (main excipient lactose monohydrate)
  Arms: biomarker treatment arm

SUMMARY:
Cough is a common symptom of respiratory medicine clinic patients, which has complex etiology and wide-ranging. Cough is usually divided into three categories by time: acute cough, subacute cough and chronic cough. Subacute has a 3~8 weeks course of disease. Its main etiology is postinfectious cough, which is mostly secondary to viral infection.Considering its overexpression in postinfectious patient, Cysteinyl leukotriene (CysLTs) plays a role in gathering eosinophils to respiratory. The level of FENO has a significant correlation with inflammatory airway eosinophils. While CysLTs overexpressed in vivo, the level of FENO may increase. Montelukast, as CysLTs-receptor-1 antagonists， plays a role of controlling airway inflammation and decrease airway high activity by suppressing the biological activity of CysLTs. It is effective in theory to therapy sub-acute cough by Montelukast, to short the course and to relieve cough symptoms as soon as possible. The aim is to research whether FENO can be used as a biomarker to optimized treatment regimen of sub-acute cough.

DETAILED DESCRIPTION:
This project is a prospective, open label, randomized and controlled trial. All subacute cough patients that met the inclusion/exclusion criteria were recruited after signing the consent form. Patients were randomized into biomarker treatment arm and standard treatment arm. Positive or negative biomarker expression was confirmed by assessing fractional concentration of exhaled NO (FENO) level, FENO<25ppb was regarded as negative and FENO≥25ppb was regarded as positive.

Patients in biomarker guided positive treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) . Patients in biomarker guided negative treatment arm were given placebo tablets(p.o., 10mg, q.d.). Patients in standard treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.).All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.

Examine results of all patients from all arms were recorded before and after the 10 day treatment. The examine recorded are FENO levels, cough symptom assessment, cough visual assessment, Leicester cough questionnaire, total white blood cell count, neutrophil blood percentage, eosinophil blood percentage. Patient cough free days after treatment and Montelukast Sodium Tablets . Follow up was carried out at the 8th week after first record of symptom and 2 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cough is the main or only clinical symptom and was persistent for 3-8 weeks
* Chest X-ray reveals no noticeable pathological changes
* ≥18 year old, regardless of gender and ethical background
* Not taking angiotensin-converting enzyme inhibitor
* Patients must join the programme voluntarily and are able to attend examination and follow-up sessions

Exclusion Criteria:

* Patients diagnosed with rhinallergosis, chronic nasosinusitis or bacterial respiratory tract infections
* Patients diagnosed with severe reportorial disease of other severe systemic disease
* Patients who are allergic to any drugs to be tested
* Patients who are non-cooperative during examination sessions or other steps of the trial
* Patients who are not able to or refuse to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Leicester cough questionnaire | 10 days

SECONDARY OUTCOMES:
cough visual assessment | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Kewu Huang, M.D., Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Morice AH, Fontana GA, Sovijarvi AR, Pistolesi M, Chung KF, Widdicombe J, O'Connell F, Geppetti P, Gronke L, De Jongste J, Belvisi M, Dicpinigaitis P, Fischer A, McGarvey L, Fokkens WJ, Kastelik J; ERS Task Force. The diagnosis and management of chronic cough. Eur Respir J. 2004 Sep;24(3):481-92. doi: 10.1183/09031936.04.00027804. No abstract available. PMID 15358710
- [Background] Kwon NH, Oh MJ, Min TH, Lee BJ, Choi DC. Causes and clinical features of subacute cough. Chest. 2006 May;129(5):1142-7. doi: 10.1378/chest.129.5.1142. PMID 16685003
- [Background] Lim KG, Mottram C. The use of fraction of exhaled nitric oxide in pulmonary practice. Chest. 2008 May;133(5):1232-42. doi: 10.1378/chest.07-1712. PMID 18460522
- [Background] McCool FD. Global physiology and pathophysiology of cough: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):48S-53S. doi: 10.1378/chest.129.1_suppl.48S. PMID 16428691
- [Background] Mita H, Turikisawa N, Yamada T, Taniguchi M. Quantification of leukotriene B4 glucuronide in human urine. Prostaglandins Other Lipid Mediat. 2007 Feb;83(1-2):42-9. doi: 10.1016/j.prostaglandins.2006.09.010. Epub 2006 Dec 5. PMID 17259071
- [Background] Ryan NM, Gibson PG. Extrathoracic airway hyperresponsiveness as a mechanism of post infectious cough: case report. Cough. 2008 Aug 4;4:7. doi: 10.1186/1745-9974-4-7. PMID 18673583
- [Background] Cho YS, Park SY, Lee CK, Lee EY, Shin JH, Yoo B, Moon HB. Enhanced cough response to hyperpnea with cold air challenge in chronic cough patients showing increased cough sensitivity to inhaled capsaicin. Allergy. 2003 Jun;58(6):486-91. doi: 10.1034/j.1398-9995.2003.00183.x. PMID 12757448
- [Background] Montuschi P, Mondino C, Koch P, Barnes PJ, Ciabattoni G. Effects of a leukotriene receptor antagonist on exhaled leukotriene E4 and prostanoids in children with asthma. J Allergy Clin Immunol. 2006 Aug;118(2):347-53. doi: 10.1016/j.jaci.2006.04.010. Epub 2006 Jul 3. PMID 16890757
- [Background] Kato A, Schleimer RP. Beyond inflammation: airway epithelial cells are at the interface of innate and adaptive immunity. Curr Opin Immunol. 2007 Dec;19(6):711-20. doi: 10.1016/j.coi.2007.08.004. Epub 2007 Oct 24. PMID 17928212
- [Background] Sato S, Saito J, Sato Y, Ishii T, Xintao W, Tanino Y, Ishida T, Munakata M. Clinical usefulness of fractional exhaled nitric oxide for diagnosing prolonged cough. Respir Med. 2008 Oct;102(10):1452-9. doi: 10.1016/j.rmed.2008.04.018. Epub 2008 Jul 9. PMID 18614345
- [Background] Seymour ML, Gilby N, Bardin PG, Fraenkel DJ, Sanderson G, Penrose JF, Holgate ST, Johnston SL, Sampson AP. Rhinovirus infection increases 5-lipoxygenase and cyclooxygenase-2 in bronchial biopsy specimens from nonatopic subjects. J Infect Dis. 2002 Feb 15;185(4):540-4. doi: 10.1086/338570. Epub 2002 Jan 31. PMID 11865407
- [Background] Gentile DA, Fireman P, Skoner DP. Elevations of local leukotriene C4 levels during viral upper respiratory tract infections. Ann Allergy Asthma Immunol. 2003 Sep;91(3):270-4. doi: 10.1016/S1081-1206(10)63529-6. PMID 14533659
- [Background] van Schaik SM, Tristram DA, Nagpal IS, Hintz KM, Welliver RC 2nd, Welliver RC. Increased production of IFN-gamma and cysteinyl leukotrienes in virus-induced wheezing. J Allergy Clin Immunol. 1999 Apr;103(4):630-6. doi: 10.1016/s0091-6749(99)70235-6. PMID 10200012
- [Background] Kim CK, Koh JY, Han TH, Kim DK, Kim BI, Koh YY. Increased levels of BAL cysteinyl leukotrienesinacute [corrected] RSV bronchiolitis. Acta Paediatr. 2006 Apr;95(4):479-85. doi: 10.1080/08035250600554268. PMID 16720498
- [Background] Payne DN, Adcock IM, Wilson NM, Oates T, Scallan M, Bush A. Relationship between exhaled nitric oxide and mucosal eosinophilic inflammation in children with difficult asthma, after treatment with oral prednisolone. Am J Respir Crit Care Med. 2001 Oct 15;164(8 Pt 1):1376-81. doi: 10.1164/ajrccm.164.8.2101145. PMID 11704581
- [Background] Berry MA, Shaw DE, Green RH, Brightling CE, Wardlaw AJ, Pavord ID. The use of exhaled nitric oxide concentration to identify eosinophilic airway inflammation: an observational study in adults with asthma. Clin Exp Allergy. 2005 Sep;35(9):1175-9. doi: 10.1111/j.1365-2222.2005.02314.x. PMID 16164444